CLINICAL TRIAL: NCT06007794
Title: Correlation Between Ultrasound-assessed Quadriceps Muscle Mass and Baseline Whole-body Densitometry Muscle Index in the Post-cancer Population (JUMP Research II)
Acronym: JUMPresearchII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL23_0368
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Post-cancer; Hematology
Keywords: post-cancer; sarcopenia; medical evaluation; muscle
MeSH Terms: conditions — Neoplasms; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JUMP group (Experimental): This study concerns adults with cancer treated with chemotherapy, radiotherapy, hormonal therapy or immunotherapy, in remission or cured. Patients took part in the dedicated post-cancer assessment day. In addition, an ultrasound of the thigh is performed to measure the size of the quadriceps on 5 different measurements.
  Interventions: Other: JUMP group

INTERVENTIONS:
Other: JUMP group — patients will have a femoral ultrasound and blood tubes in addition to the blood sample taken as part of the treatment

SUMMARY:
Therapeutic advances in oncology have transformed the prognosis of cancer patients, placing a significant number of them either in a context of recovery or in prolonged remission close to a chronic disease. Thus, the reconquest of a life after cancer becomes possible but raises many challenges for the patient, his entourage, the medical profession and our society. One of the major challenges is the detection and management of treatment side effects for all patients. In addition to the standard organic assessment (glycaemia, creatinine, liver test, blood count), we are mainly interested in muscle deconditioning and cognitive impairment, which are particularly disturbed in these populations. After the evaluation day, patients are referred to the most appropriate structures (Adapted physical activity, sports for health, and rehabilitation at Henry Gabriel Hospital).

JUMP research is part of axis 2 of the 2021-2030 cancer plan: "Limiting sequelae and improving quality of life", through sheets 1 (research) / 6 (access and quality) / 7 (prevention). This leads to the concrete implementation on the territory of adapted care channels in the city: medical structure, physiotherapy, Adapted Physical Activity (APA) structures, associative structures; which makes it possible to develop and strengthen the city-hospital link. Finally, it allows the patient to take ownership and get involved in the project, allowing in the future to make them truly active in they care and to advise and motivate their peers.

This non-interventional research is classified as "research involving human subjects", class 3 .

The objective of this research is to evaluate the impact of cancer on the musculoskeletal system and to test ultrasound as a clinical examination for the detection of sarcopenia in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 to 74 years
* localization of the primitive: breast, lung, melanoma, testicle, bladder, kidney, ovary, colon and pancreas, hemopathy
* patient who benefited from the post-cancer assessment day

Exclusion Criteria:

* Active cancer (relapse or new cancer)
* Pregnant or breastfeeding women
* Major cognitive impairment making comprehension and exercise difficult
* Amputation of both lower limbs (for ultrasound)
* Difficulty understanding oral and written French
* Adults under legal protection (guardianship, curatorship or safeguard of justice)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2029-02-10 (Estimated); Study Completion 2029-05-10 (Estimated)

PRIMARY OUTCOMES:
Analyze the correlation between muscle mass (thickness) of the quadriceps (rectus femoris) assessed in axial sections by ultrasound and the reference muscle mass index (Appendicular Lean Mass (ALM)/height²) assessed by DEXA | through study completion, an average of 9 years
  Analyze the correlation between muscle mass (thickness) of the quadriceps (rectus femoris) assessed in axial sections by ultrasound and the reference muscle mass index (Appendicular Lean Mass (ALM)/height²) assessed by DEXA Mean thickness of the quadriceps (straight femoris) measured by ultrasound compared to the Appendicular Lean Mass/size² in DEXA

SECONDARY OUTCOMES:
Correlation between the ultrasound muscle indexes and the scannographic index of the paravertebral muscles (SMI L3, T12 and T7, studied by IA) | through study completion, an average of 9 years
  Evaluation of the section surface of the rectus femoris in ultrasound, of the adipose infiltration index of the rectus femoris on ultrasound and of the Skeletal Muscle Index (SMI) L3, T12 and T7 in CT (gold standard)
Correlation between ultrasound muscle indices and muscle functional tests | through study completion, an average of 9 years
  Calculation of Functional Indices and questionnaire scores: grip strength, TM6, 30-second sit-to-stand test, SARC-F and IPAQ
Correlation between muscle biological markers (irisin, myostatin, FGF19, TGFb, decarboxylated osteocalcin, microRNA) and the diagnosis of sarcopenia (according to EWSGOP 2019 and BAUMGARTNER) | through study completion, an average of 9 years
  Serum biomarker assays: myostatin, irisin, micro-RNA, osteocalcin, FGF19 and diagnosis of sarcopenia assessed according to Baumgartner and to to EWSGOP 2019 definitions
Correlation between muscle biological markers (irisin, myostatin, FGF19, TGFb, decarboxylated osteocalcin, microRNA) and ultrasound, densitometric, scannographic and functional parameters | through study completion, an average of 9 years
  Serum biomarker assays: myostatin, irisin, micro-RNA, osteocalcin, FGF19, interpretation of images (ultrasound, densitometry, scanner) and results of functional tests
Reproducibility of muscle ultrasound, in a subgroup of patients, inter-observer (n=10 patients) | through study completion, an average of 9 years
  ICC of the thickness of the quadriceps, of its cross-sectional area interobserver (subpopulation of 10 patients)
Reproducibility of muscle ultrasound, in a subgroup of patients, intra-observer (n=10 patients). | through study completion, an average of 9 years
  ICC of the thickness of the quadriceps, its cross-sectional area intraobserver (subpopulation of 10 patients)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, rhumatologie, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No